CLINICAL TRIAL: NCT00408538
Title: A Phase 1 Randomized, Blinded, Placebo-Controlled Safety and Acceptability Study of the UC-781 Vaginal Microbicide Gel Formulation Applied Rectally in HIV-1 Seronegative Adults
Brief Title: Safety and Acceptability Study of the UC-781 Microbicide Gel Applied Rectally
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); CONRAD (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: U19-AI060614:P4 Aim 1; 06-04-043; U19AI060614 (NIH)
Record Dates: First submitted 2006-12-06; First posted 2006-12-07 (Estimated); Last update posted 2009-05-04 (Estimated); Status verified 2009-05

CONDITIONS: HIV Infections
Keywords: Microbicide; HIV; Prevention; Rectal; HIV Prevention
MeSH Terms: conditions — HIV Infections

INTERVENTIONS:
Drug: UC-781 microbicide gel (0.1% and 0.25%)
Drug: placebo

SUMMARY:
This study is the first to try this product in the rectum of humans. This study is only to find out if the gel is safe for use in the rectum, not to see if the gel works. Information gathered from this study will help investigators decide whether this gel is safe enough to move onto the next phase of studies.

Information gathered from this study will also help investigators determine what participants did and did not like about the product and what types of products people might want to use in the future. Currently condoms and abstinence are the only methods proven to prevent the spread of HIV sexually.

DETAILED DESCRIPTION:
The purpose of this study is to obtain preliminary data on the safety and acceptability of UC-781 vaginal microbicide gel (0.1% and 0.25%) versus placebo when rectally administered in HIV-1 seronegative adults.

Participants will enter a screening period, which includes Visit 1 and if necessary a medication washout period.

Subjects who are deemed eligible after this screening period will return for a baseline evaluation (Visit 2), including clinical evaluation and mucosal specimen collection, as well as the Baseline Behavioral Questionnaire (BBQ). The BBQ will be administered by Computer Assisted Self-Interview (CASI). Subjects may complete the web-based CASI in the privacy of their own home. If a subject does not have access to the Internet, prefers to complete the BBQ at the study site, or requires assistance in using the CASI, he or she will be accommodated at the study site.

After completing Visits 1 and 2, eligible subjects will be randomized to one of three groups: 0.1% UC-781 gel, 0.25% UC-781 gel, or a placebo gel (12 per group). A subset of 9 subjects (3 from each group) will also participate in a pK sub-study, which will include 6 timepoints (Visit 3- pre, 0.25 hr, 2 hr, 4 hr, Visit 3A- 24 hr, and Visit 5- 1 day post-QD dose). During randomization, study staff will be notified if the participant is randomized to the pK substudy.

This study will involve 2 stages of treatment. Each treatment stage is independent of the other. This study aims to examine the effects of 2 different dosing regimens, NOT cumulative safety over the both stages.

Once randomized, subjects will return to the clinic (Visit 3), where a single dose of the study gel (Treatment Stage 1) will be administered followed by clinical evaluation, including flexible sigmoidoscopy, and sample collection.

Subjects will return to the clinic for Treatment Stage 2 Clearance (Visit 4), in the week prior to beginning Treatment Stage 2. If given clearance, the subject may begin Treatment Stage 2.

In Treatment Stage 2, subjects will begin to self-administer once daily outpatient doses of the study gel for 7 days. After completion of Stage 2 the subject will complete a Product Acceptability Questionnaire (PAQ) by CASI and return to clinic for evaluation and specimen collection (Visit 5).

After completion of Visit 5, subjects will be contacted by an interviewer to complete an in-depth phone interview regarding product acceptability.

ELIGIBILITY:
Inclusion Criteria:

Men who meet the following 10 criteria and women who meet the following 12 criteria are eligible for inclusion in the study:

1. ≥ Age of 18
2. HIV-1 status antibody negative as documented at screening
3. Understands and agrees to local STI reporting requirements
4. Able and willing to communicate in English
5. Able and willing to provide written informed consent
6. Able and willing to provide adequate information for locator purposes
7. Availability to return for all study visits
8. A history of consensual RAI at least once in lifetime:

   * Required to assure that subjects have a context for the acceptability assessments
9. Willing to abstain from insertion of anything per rectum other than the study gel for the 1 week prior to treatment, 1 week prior each flexible sigmoidoscopy (i.e., during week of study gel use), and 1 week after each flexible sigmoidoscopy
10. Must agree to use condoms for the duration of the study

    In addition to the criteria listed above, female participants must meet the following criteria:
11. Negative pregnancy test
12. Post-menopausal or using an acceptable form of contraception (e.g. barrier method, IUD, hormonal contraception, surgical sterilization, or vasectomization of male partner). If the female subject has female partners only, the method of contraception will be noted as a barrier method in the study documentation.

Exclusion Criteria:

Individuals who meet any of the following criteria at screening will be excluded from the study:

1. HIV positive at baseline
2. History of inflammatory bowel disease
3. Active inflammatory condition of the GI tract at baseline
4. Active rectal infection at baseline
5. ≥ Grade 2 laboratory abnormality (≥ Grade 1 potassium, magnesium, chloride, sodium, and calcium) at baseline
6. History of an underlying cardiac arrhythmia or renal disease that may be exacerbated by electrolyte abnormalities
7. History of severe or recent cardiac or pulmonary event
8. History of a large aortic aneurysm
9. History of significant gastrointestinal bleeding
10. Allergy to methylparaben, propylparaben, sorbic acid
11. History of alcoholism or IV drug abuse
12. Unwillingness to refrain from chronic use of aspirin and NSAIDs
13. Use of warfarin or heparin
14. Use of systemic immunomodulatory medications within 4 weeks of Visit 2
15. Use of rectally administered medications, with the exception of over-the-counter enemas, within 4 weeks of Visit 2
16. Use of product containing nonoxyl-9 rectally within 4 weeks of Visit 2
17. Use of any investigational products within 4 weeks of Visit 2
18. Any other clinical condition or prior therapy that, in the opinion of the investigator, would make the patient unsuitable for the study or unable to comply with the study requirements. Such conditions may include, but are not limited to, current or recent history of severe, progressive, or uncontrolled renal, hepatic, hematological, gastrointestinal, endocrine, pulmonary, neurological, or cerebral disease.

    In addition to the criteria listed above, female participants will be excluded if the meet any of the following criteria:
19. Pregnancy
20. Breastfeeding
21. Female of child-bearing potential unwilling to use acceptable form of contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2006-12; Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Frequency of ≥ Grade 2 adverse events
Acceptability assessments

SECONDARY OUTCOMES:
Epithelial sloughing
Histopathology
Microflora
Mucosal mononuclear cell phenotype
Mucosal cytokine profile
Mucosal immunoglobulins
Fecal calprotectin
Explants- Mucosal cytokine profile and susceptibility to HIV infection

CONTACTS AND LOCATIONS:
Locations (1):
- UCLA Center for HIV Prevention Research, Los Angeles, California, United States

REFERENCES:
- [Derived] Richardson-Harman N, Mauck C, McGowan I, Anton P. Dose-response relationship between tissue concentrations of UC781 and explant infectibility with HIV type 1 in the RMP-01 rectal safety study. AIDS Res Hum Retroviruses. 2012 Nov;28(11):1422-33. doi: 10.1089/AID.2012.0073. Epub 2012 Sep 20. PMID 22900504
- [Derived] Anton PA, Saunders T, Elliott J, Khanukhova E, Dennis R, Adler A, Cortina G, Tanner K, Boscardin J, Cumberland WG, Zhou Y, Ventuneac A, Carballo-Dieguez A, Rabe L, McCormick T, Gabelnick H, Mauck C, McGowan I. First phase 1 double-blind, placebo-controlled, randomized rectal microbicide trial using UC781 gel with a novel index of ex vivo efficacy. PLoS One. 2011;6(9):e23243. doi: 10.1371/journal.pone.0023243. Epub 2011 Sep 28. PMID 21969851